CLINICAL TRIAL: NCT05229614
Title: Immune Checkpoint Inhibitors and Carbon iON Radiotherapy In Solid Cancers With Stable Disease
Brief Title: Immunotherapy and Carbon Ion Radiotherapy In Solid Cancers With Stable Disease
Acronym: ICONIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Italy (Unknown); Fondazione IRCCS Policlinico San Matteo, Pavia, Italy (Unknown); GSI Helmholtzzentrum für Schwerionenforschung GmbH, Darmstadt, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNAO 44 2021 C
Record Dates: First submitted 2022-01-10; First posted 2022-02-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Melanoma; Urothelial Carcinoma
Keywords: Hadrontherapy; CIRT; Immunotherapy; NSCLC; HNSCC; Melanoma; Urothelial
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Melanoma; Carcinoma, Transitional Cell | interventions — Heavy Ion Radiotherapy; Immunotherapy; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patient with solid cancer (NSCLC, HNSCC, melanoma, urothelial carcinoma) and a stable disease will be enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Solid cancers with stable disease (Experimental): Only cancer patients under treatment with pembrolizumab monotherapy, administered within clinical practice and according to the Italian Drug Regulatory Agency (Agenzia Italiana del Farmaco, AIFA), will be enrolled.
  Patients diagnosed with NSCLC, HNSCC, melanoma and urothelial carcinoma will be eligible for the study.
  Interventions: Radiation: Carbon Ion Therapy; Drug: Immunotherapy (Pembrolizumab)

INTERVENTIONS:
Radiation: Carbon Ion Therapy — After confirming the disease stability and upon patient inclusion in the study, hypofractionated carbon ion boost will be administered to one site of disease previously untreated. Patient will be irradiated to a single lesion with a total dose of 24 Gy[RBE], 8 Gy[RBE]/fraction, one fraction/day, for 3 days.
Drug: Immunotherapy (Pembrolizumab) — Only cancer patients under treatment with pembrolizumab monotherapy, administered within clinical practice and according to the Italian Drug Regulatory Agency (Agenzia Italiana del Farmaco, AIFA), will be enrolled.
  Other Names: Pembrolizumab

SUMMARY:
Immunotherapy has become the standard of care in different advanced malignancies. Its effectiveness in the palliative setting was demonstrated by several phase III trials. However, the response rate varies according to the cancer under study and to the line of treatment. A potential way to improve the activity of single agent immune checkpoint inhibitors (ICIs) is to enhance the clinical response through further antitumor agents, including radiotherapy. Studies showed that carbon ions may lead to a broader immunogenic response; for their dosimetric characteristics it is possible to reduce integral dose sparing immune cells to direct and sustain a tumor specific immune response.

Considering the available preclinical and clinical evidence together, the goal of this study is to explore the feasibility and the clinical activity of adding carbon ion radiotherapy (CIRT), employed with a fractionation strategy comparable to stereotactic body radiation, to ICIs in advanced malignancies where immunotherapy is currently the standard of care.

DETAILED DESCRIPTION:
This is a multicenter, open label, non-randomized phase II clinical trial aiming to assess the feasibility and the clinical activity of adding CIRT to ICIs in cancer patients that have obtained a disease stability (SD) with pembrolizumab administered as per standard of care. At study entry, hypofractionated CIRT will be delivered to one measurable lesion previously untreated with local approaches.CIRT will be performed at Fondazione CNAO, Pavia

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Histologic confirmation of malignancies under treatment with single agent anti-PD1/PDL1 immunotherapy per clinical practice (see cohort specific inclusion criteria) with immune checkpoint inhibitors approved by Italian national drug regulatory agencies (Agenzia Italiana del Farmaco, AIFA)
3. Having a disease stability as assessed by AIFA monitoring sheet
4. Presence of at least 2 measurable target lesions, of which at least one to be followed up as per RECIST and one suitable for CIRT
5. Willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
6. Females and males, 18 years of age or older (no upper limit for age)
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
8. Subjects must have measurable disease by CT or MRI per RECIST 1.1

Exclusion Criteria:

1. Patients treated with chemo-immunotherapy associations
2. Patients treated with immunotherapy combinations (e.g. subjects treated with anti-CTLA4 + anti-PD1/PDL1 are excluded)
3. Patients receiving immunotherapy within clinical trials
4. Patients receiving off-label immunotherapy or within expanded access programs or as compassionate use
5. Patients with high tumor burden defined as > 10 lesions and/or sum of diameters > 19 cm
6. Patients with distant metastases only located in the CNS are excluded
7. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
8. Patients with autoimmune diseases (ADs), including local and systemic collagen-vascular (CVD) and inflammatory bowel diseases (IBD)
9. Previous RT, regardless of energy, on the metastatic site selected to be irradiated.
10. Any immune-related CTCAE grade 4 adverse event, before study entry
11. Any CTCAE grade ≥3 immune-related adverse event observed within 3 weeks prior to CIRT start
12. Presence of metal prostheses or any other condition to prevent adequate imaging for identification of the target volume and calculation of the dose
13. Loco-regional conditions not allowing hadron therapy (e.g. active infections in RT target region)
14. Prisoners or subjects who are involuntarily incarcerated
15. Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness (e.g. infectious disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate assessed by RECIST V1.1 | At least 8 weeks
  To estimate the effect, in terms of clinical response, of immunotherapy associating carbon ion treatment (CIRT) in the palliative setting across different malignancies, for which immunotherapy is currently the standard of care. Objective response rate (ORR) will be evaluated after CIRT administrated during immunotherapy maintenance in patients with stable disease. ORR will be assessed in the whole population according to RECIST v1.1. The proportion of ORR will be estimated within each disease.

SECONDARY OUTCOMES:
Treatment-related adverse events assessed by CTCAE V5.0 | At least 8 weeks
  To describe the safety profile of the association of carbon ion radiation therapy and systemic immunotherapy in the palliative setting across different malignancies, for which immunotherapy is currently the standard of care. Treatment-related adverse events will be evaluated according to CTCAE version 5.0.
Efficacy in terms of survival | At least 8 weeks
  To estimate the effect, in terms of survival, of immunotherapy with the association of carbon ion radiation treatment in the palliative setting across different malignancies, for which immunotherapy is currently the standard of care.
  Progression-Free Survival (PFS) will be calculated as the time between the start date of immunotherapy associated with carbon ion and the progression of disease, or death or last-follow-up. PFS will be estimated, within each malignancy, by Kaplan-Meier product limit method.
  Overall survival (OS) will be calculated as the time between the start date of immunotherapy associated with carbon ion and the death for any cause or last follow-up. OS will be estimated, within each malignancy, by Kaplan-Meier product limit method.

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Vitolo, MD, Principal Investigator — Fondazione CNAO
Locations (4):
- GSI Helmholtzzentrum für Schwerionenforschung GmbH, Darmstadt, Germany
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - National Center for Oncological Hadrontherapy (CNAO), Pavia
  - Fondazione IRCCS Policlinico San Matteo, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Dewan MZ, Galloway AE, Kawashima N, Dewyngaert JK, Babb JS, Formenti SC, Demaria S. Fractionated but not single-dose radiotherapy induces an immune-mediated abscopal effect when combined with anti-CTLA-4 antibody. Clin Cancer Res. 2009 Sep 1;15(17):5379-88. doi: 10.1158/1078-0432.CCR-09-0265. Epub 2009 Aug 25. PMID 19706802
- [Background] Durante M, Paganetti H. Nuclear physics in particle therapy: a review. Rep Prog Phys. 2016 Sep;79(9):096702. doi: 10.1088/0034-4885/79/9/096702. Epub 2016 Aug 19. PMID 27540827
- [Background] Deng L, Liang H, Xu M, Yang X, Burnette B, Arina A, Li XD, Mauceri H, Beckett M, Darga T, Huang X, Gajewski TF, Chen ZJ, Fu YX, Weichselbaum RR. STING-Dependent Cytosolic DNA Sensing Promotes Radiation-Induced Type I Interferon-Dependent Antitumor Immunity in Immunogenic Tumors. Immunity. 2014 Nov 20;41(5):843-52. doi: 10.1016/j.immuni.2014.10.019. Epub 2014 Nov 6. PMID 25517616
- [Background] Vanpouille-Box C, Alard A, Aryankalayil MJ, Sarfraz Y, Diamond JM, Schneider RJ, Inghirami G, Coleman CN, Formenti SC, Demaria S. DNA exonuclease Trex1 regulates radiotherapy-induced tumour immunogenicity. Nat Commun. 2017 Jun 9;8:15618. doi: 10.1038/ncomms15618. PMID 28598415
- [Background] Deng L, Liang H, Burnette B, Beckett M, Darga T, Weichselbaum RR, Fu YX. Irradiation and anti-PD-L1 treatment synergistically promote antitumor immunity in mice. J Clin Invest. 2014 Feb;124(2):687-95. doi: 10.1172/JCI67313. Epub 2014 Jan 2. PMID 24382348
- [Background] Antonioli L, Blandizzi C, Pacher P, Hasko G. Immunity, inflammation and cancer: a leading role for adenosine. Nat Rev Cancer. 2013 Dec;13(12):842-57. doi: 10.1038/nrc3613. Epub 2013 Nov 14. PMID 24226193
- [Background] Golden EB, Demaria S, Schiff PB, Chachoua A, Formenti SC. An abscopal response to radiation and ipilimumab in a patient with metastatic non-small cell lung cancer. Cancer Immunol Res. 2013 Dec;1(6):365-72. doi: 10.1158/2326-6066.CIR-13-0115. PMID 24563870
- [Background] Dovedi SJ, Adlard AL, Lipowska-Bhalla G, McKenna C, Jones S, Cheadle EJ, Stratford IJ, Poon E, Morrow M, Stewart R, Jones H, Wilkinson RW, Honeychurch J, Illidge TM. Acquired resistance to fractionated radiotherapy can be overcome by concurrent PD-L1 blockade. Cancer Res. 2014 Oct 1;74(19):5458-68. doi: 10.1158/0008-5472.CAN-14-1258. PMID 25274032
- [Background] Tang C, Welsh JW, de Groot P, Massarelli E, Chang JY, Hess KR, Basu S, Curran MA, Cabanillas ME, Subbiah V, Fu S, Tsimberidou AM, Karp D, Gomez DR, Diab A, Komaki R, Heymach JV, Sharma P, Naing A, Hong DS. Ipilimumab with Stereotactic Ablative Radiation Therapy: Phase I Results and Immunologic Correlates from Peripheral T Cells. Clin Cancer Res. 2017 Mar 15;23(6):1388-1396. doi: 10.1158/1078-0432.CCR-16-1432. Epub 2016 Sep 20. PMID 27649551
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Derived] Cavalieri S, Vitolo V, Barcellini A, Ronchi S, Facoetti A, Campo C, Klersy C, Molinelli S, Agustoni F, Ferretti VV, Silvestri A, Platania M, Del Vecchio M, Durante M, Helm A, Fournier C, Braud F, Pedrazzoli P, Orlandi E, Licitra L. Immune checkpoint inhibitors and Carbon iON radiotherapy In solid Cancers with stable disease (ICONIC). Future Oncol. 2023 Jan;19(3):193-203. doi: 10.2217/fon-2022-0503. Epub 2023 Mar 28. PMID 36974574